CLINICAL TRIAL: NCT01245114
Title: Tübingen High Altitude Ophthalmology Study (THAO)
Brief Title: Tübingen High Altitude Ophthalmology Study
Acronym: THAO
Status: Completed | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Prof. Florian Gekeler, Eye Hospital, University Hospital Tübingen, Germany
Other Study IDs: THAO
Record Dates: First submitted 2010-11-19; First posted 2010-11-22 (Estimated); Last update posted 2010-12-03 (Estimated); Status verified 2010-07

CONDITIONS: Altitude; Hypoxia
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Tuebingen High Altitude Ophthalmology Study to investigate the effects of high altitude on retinal structure and function as well as anterior chamber in regard to acute mountain sickness.

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects, non-smokers, physical fitness,

Exclusion Criteria:

* ocular pathologies, ascent above 2000m 2 weeks prior to study and 2 weeks before post-examination

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy volunteers
Sampling Method: Probability Sample
Dates: Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Florian Gekeler, MD, Study Director — Eye Hospital, University of Tübingen, Germany; Gabriel Willmann, MD, Principal Investigator — Eye Hospital, University of Tübingen, Germany
Locations (1):
- Eye Hospital, University of Tübingen, Tübingen, Baden-Wurttemberg, Germany